CLINICAL TRIAL: NCT03274609
Title: CT-controlled Advanced Navigation Techniques for Transbronchial Pulmonary Lesion Access; Evaluation of Augmented Fluoroscopy Bronchoscopic Navigation Based Diagnostic Yield
Acronym: CONTROL-A
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL63109.091.17
Record Dates: First submitted 2017-08-17; First posted 2017-09-07 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2018-04

CONDITIONS: Lung Cancer
Keywords: Lung diseases; cancer; Interventional pulmonology; peripheral nodule
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — biopsies of peripheral nodules
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Suspected lung cancer: * Patients referred as part of a first diagnostic evaluation of newly detected pulmonary lesion(s) or when an indication for an invasive diagnostic procedure is found during follow-up of earlier detected pulmonary lesion.
  * Patients identified during per protocol CT imaging follow-up of known lesions when growth of the lesion is found and an indication for biopsy is determined by the treating physician and/or multidisciplinary board.
  * Patients identified when referred for surgical biopsy in case of nodule location inaccessible for CT-guided TTNA.
  These will be subjected to a combined approach of modalities with the main intervention being augmented fluoroscopy guided virtual navigation.)
  Interventions: Combination Product: Augmented fluoroscopy

INTERVENTIONS:
Combination Product: Augmented fluoroscopy — Augmented fluoroscopy based virtual navigation combined with use of radial EBUS probe and Rapid On Site Evaluation of Histology for diagnosis of peripheral pulmonary nodules.Controlled by cone beam CT.

SUMMARY:
In this exploratory adaptive clinical trial the investigators will examine the diagnostic yield of a combination of commercially available imaging and navigation techniques for reaching peripheral lung lesions. The two investigated techniques will herein be the rEBUS imaging modality combined with augmented fluoroscopy based virtual bronchoscopy navigation. Confirmation of reaching the lung lesion will be by means of CT (fluoroscopic) imaging. Rapid On-Site Evaluation (ROSE) of cytopathology will be used for obtaing a per-procedural outcome on tissue biopsy representativeness. The study will replace the current conventional standard TBB procedure (fluoroscopy and rEBUS guided bronchoscopy) in the endoscopy suite. Consecutive patients will be included on the MITeC hybrid operating room (needed to monitor patient safety and CT availability). All data will be prospectively collected. In case tissue biopsy is found to be malignant or benign, it will be termed representative. In case tissue biopsy is found to be non-representative (=blood, anatomical lung tissue, unreachable), conventional follow-up of CT guided TTNA, follow-up monitoring and/or surgical biopsy will serve as golden standard for obtaining tissue diagnosis. For verification of reaching the target lesion, another study parameter of interest, (cb)CT imaging will be performed for verification that instruments are within the nodule (per-procedurally available).

DETAILED DESCRIPTION:
Lung cancer is one of the leading most frequent types of cancer and is the most lethal malignancy in the Netherlands. Mortality is high due to its advanced stage disease at diagnosis. To improve survival current guidelines are moving towards CT-screening of the high risk population. These CT-scans detect numerous nodules and rapidly increase the demand for minimal invasive accurate and safe diagnostic procedures.

The historically available and current first diagnostic procedure in the work-up of PPLs is fluoroscopy guided Trans Bronchial Biopsy (TBB) despite its low pooled yield of 31.1%. When the above transbronchial technique does not provide an unambiguous outcome, an additional and more invasive diagnostic work-up remains indicated. To exclude the possibility of missing malignancies, trans thoracic needle aspiration is first indicated. If deemed inaccessible, surgical biopsy may be alternatively indicated depending on patient risk of malignancy. Ideally, a transbronchial approach having high diagnostic accuracy would overcome the need of this sequential increasingly invasive diagnostic and consecutive treatment approach. Newer pilot studies now hypothesize that combining multiple new endobronchial modalities might provide a solution in preventing more invasive additional diagnostic staging, reporting diagnostic yields exceeding 70%. When an accurate and certain transbronchial diagnosis by combining multiple techniques can indeed be provided. We will study a combination of new advanced modalities for diagnosis of peripheral nodules endobronchially. The aim of this study is to determine diagnostic yield, cost-effectiveness, safety, and, to collect data for developing diagnostic algorithms to further cost-effectively increase yield, reduce complication rate and determine a future platform for clinical implementation.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* ASA physical status 1-3.
* Age 18 years or older.
* A pulmonary lesion (i.e. a focal, rounded opacity mostly surrounded by aerated lung or a ground glass opacity or part- or sub-solid lesion) with an indication for diagnostic evaluation following current clinical guidelines and/or as decided by multi-disciplinary team consultation.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Bleeding disorders.
* Less than 18 years old.
* Contra-indication for temporary interruption of the use of anticoagulant therapy (acenocoumarol, warfarin, therapeutic dose of low molecular weight heparines, clopidrogel, analogs, or, NOAC's).
* Known allergy for lidocaine.
* Uncontrolled pulmonary hypertension.
* Recent and/or uncontrolled cardiac disease.
* Compromised upper airway (e.g. concomitant head and neck cancer or central airway stenosis for any reason such that endobronchial access is considered unsafe).
* ASA classification greater than or equal to 4 (unfit for performing non-surgical biopsy).
* Pregnancy.
* Inability to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients diagnosed with peripheral pulmonary lesion(s) and an indication to obtain a tissue sample(s) following current conventional procedure work-up. In all patients, preprocedural imaging (including CT and/or PET-CT findings) following conventional work-up is available. Case selection for the clinical indication to perform a peripheral pulmonary biopsy (non-surgical and/or surgical) will follow current local clinical practice, multidisciplinary tumor board decisions and is in accordance to the latest British Thoracic Society guidelines (British Thoracic Society Pulmonary Nodule Guideline Development Group, 2015). Patients are eligible after informed consent is obtained and when direct contra-indications for the endobronchial procedure are absent.
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
number of patients with an adequate diagnosis (=diagnostic yield) | 0-12 months
  diagnosis will consist of benign, malign or non-representative (=blood, anatomical lung tissue, unreachable)

SECONDARY OUTCOMES:
number of patients with (S)AE's related to the procedure | 0-12 months
  minor bleeding and pneumothoraces are reported
cost-effectiveness | 0-12 months
  the study procedures will be compared against the conventional diagnostic TBB work-up
radiation exposure | 0-12 months
  compared against conventional TBB and consecutive TTNA procedure

CONTACTS AND LOCATIONS:
Overall Officials: Linda Garms, Study Chair — Study coordinator; Erik van der Heijden, MD PhD, Principal Investigator — Pulmonary diseases; Roel Verhoeven, Msc, Study Chair — Pulmonary diseases / Radiology
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No